CLINICAL TRIAL: NCT04991233
Title: The Effectiveness and Safety of Endoscopic Evacuation Versus Suboccipital Craniotomy in the Treatment of Spontaneous Intracerebellar Hemorrhage (SCH) -a Randomized Control Trial.
Brief Title: The Treatment Effect of Endoscopic Evacuation Versus Suboccipital Craniotomy for Spontaneous Intracerebellar Hemorrhage.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDSJWK-SCH-EESC-RCT
Record Dates: First submitted 2021-04-07; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Posterior Fossa Hemorrhage
Keywords: Posterior Fossa Hemorrhage; Endoscopic Surgery; Suboccipital Craniotomy; Treatment Outcome
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The grouping was blind to the investigators performing the follow-up and the statistical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic surgery (Experimental): Endoscopic surgery group
  Interventions: Procedure: Endoscopic surgery
- Suboccipital craniotomy surgery (Active Comparator): Suboccipital craniotomy surgery group
  Interventions: Procedure: Suboccipital craniotomy surgery

INTERVENTIONS:
Procedure: Endoscopic surgery — The endoscopic surgery will be conducted to evacuate the hemorrhage within 24 hours after SCH.
  Arms: Endoscopic surgery
Procedure: Suboccipital craniotomy surgery — The suboccipital craniotomy surgery will be conducted to evacuate the hemorrhage within 24 hours after SCH.
  Arms: Suboccipital craniotomy surgery

SUMMARY:
The purpose of the present study is to compare the effectiveness and safety of two surgery evacuation methods (endoscopic surgery and suboccipital craniotomy) in the treatment of acute spontaneous cerebellar hemorrhage (SCH). A multi-center randomized control trial will be conducted. Patients with an initial GCS score of 5-14 will be screened and enrolled in the first 24 hours after SCH.

DETAILED DESCRIPTION:
Spontaneous cerebellar hemorrhage (SCH) accounts for about 9-10% of all ICH cases, with a mortality rate of 20-50%. Suboccipital craniotomy was the traditional surgery method in the treatment of SCH. Minimally invasive techniques, including endoscopic evacuation and minimally invasive catheter (MIC) evacuation, have been used for the treatment of SCH) in recent years. However, credible evidence is still needed to validate the effects of these techniques. The treatment effect of endoscopic evacuation and MIC evacuation was compared in our previous study, results showed that the endoscopic evacuation significantly decreased the 6-month mortality of SCH patients. Thus endoscopic evacuation might be a safer and more effective option in the treatment of SCH. Therefore, in the current study, a multi-center randomized control trial will be conducted to compare the effectiveness and safety of endoscopic surgery and suboccipital craniotomy in the treatment of acute SCH. A multi-center randomized control trial will be conducted. Patients with an initial GCS score of 5-14 will be screened according to the selecting criteria. The enrolled patients will undertake the surgery within the first 24 hours after SCH. The primary outcome is the 30-day mortality rate. And the secondary outcomes including the 6-month mRS, the incidence of adverse events within 30-day, the hematoma clearance rate, the residual hematoma volume on postoperative day 1/3/7, and the perihematoma edema volume on postoperative day 1/3/7.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years old;
2. Cerebellar hemorrhage was confirmed by computed tomography (CT) scans;
3. The hematoma was > 3 cm in diameter or the hematoma volume was > 10ml or the hemorrhage is associated with brainstem compression or hydrocephalus;
4. The randomization can be conducted within 24 hours;
5. GCS score at randomization was 5-14;
6. mRS was 0-1 before onset;
7. The systolic pressure was controlled below 180 mmHg before randomization;
8. Informed consent was obtained from the patient and his legal representative.

Exclusion Criteria:

1. Coexistent intracranial bleeding from other sites;
2. Brain herniation before randomization;
3. Bleeding caused by other reasons such as aneurysm, arteriovenous malformation, trauma, and tumor; hemorrhage secondary to large cerebral infarction, beta-amyloid degeneration disease, or coagulation dysfunction; coexistent aneurysm, arteriovenous malformation, brain trauma, brain tumors, large area cerebral infarction, beta-amyloid degeneration disease, or serious blood coagulation disorders;
4. A history of cerebral hemorrhage within 1 year;
5. A history of intracranial surgery or hemorrhagic disease (intracerebral hemorrhage, subarachnoid hemorrhage, subdural or epidural hemorrhage) within the last 30 days;
6. Hemoglobin < 100g/L, hematocrit < 25%, platelet count <100*10^9/L;
7. Warfarin, dabigatran, rivaroxaban, and other anticoagulant drugs were given within one week before enrollment, and the INR was > 1.4;
8. Aspirin, clopidogrel, ticagrelor, and other antiplatelet drugs were given within one week before enrollment, and the inhibition rate of AA-dependent pathway > 50%，inhibition rate of ADP-dependent pathway > 30%;
9. Long-term anticoagulation and antiplatelet therapy is needed;
10. A history of internal bleeding that is not completely controlled, such as gastrointestinal bleeding, genitourinary bleeding, respiratory bleeding;
11. Myocardial infarction within 30 days;
12. Patients with high risks of embolization (a history of mechanical heart valve implantation, left ventricular thrombosis, mitral stenosis with atrial fibrillation, acute pericarditis, or subacute bacterial endocarditis); atrial fibrillation without mitral stenosis is acceptable;
13. Severely impaired liver function (ALT > 3 times the normal upper limit, or AST > 3 times the normal upper limit); severely impaired renal function (glomerular filtration rate < 30ml/min/1.73m2);
14. Hypertension could not be effectively controlled before randomization (systolic blood pressure ≥ 180 mmHg);
15. Patients cannot complete the follow-up due to Alzheimer's disease or mental illness;
16. Coexistent serious diseases of the respiratory, circulatory, digestive, urogenital, endocrine, immune, and blood systems that are likely to interfere with the results;
17. Patients with current drug/alcohol abuse or dependence, or expected to have poor compliance and difficult to complete the follow-up;
18. Allergic to the drugs or instruments used in surgery;
19. Patients with surgery contraindications, or the other factors that may preclude implementation of the study protocol;
20. Pregnant or lactating women;
21. Life expectancy < 12 months due to any advanced stage of disease;
22. Patient is participating in other clinical trials;
23. The legal guardian of the patient is unwilling to sign the written informed consent;
24. Assessed unsuitable for inclusion by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mortality Rate | Within 30 days after SCH
  The mortality rate in each group at 30 days after SCH.

SECONDARY OUTCOMES:
mRS Score | Within 6 months after SCH
  The mortality rate in each group at 6 months after SCH.
Adverse Events | Within 30 days after SCH
  The Incidence of adverse events within 30 days after SCH.
Residual Hematoma Volume | Within 7 days after SCH
  The residual hematoma volume on postoperative day 1, day 3 and day 7.
Perihematoma Edema Volume | Within 7 days after SCH
  The perihematoma edema volume on postoperative day 1, day 3 and day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qu, M.D Ph.D, Study Chair — Tang-Du Hospital; Wei Guo, M.D Ph.D, Study Director — Tang-Du Hospital
Locations (1):
- Tandu Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li L, Liu H, Luo J, Tan Z, Gao J, Wang P, Jing W, Fan R, Zhang X, Guo H, Bai H, Cui W, Wu X, Qu Y, Guo W. Comparison of Long-Term Outcomes of Endoscopic and Minimally Invasive Catheter Evacuation for the Treatment of Spontaneous Cerebellar Hemorrhage. Transl Stroke Res. 2021 Feb;12(1):57-64. doi: 10.1007/s12975-020-00827-8. Epub 2020 Jul 4. PMID 32623579
- [Background] Heros RC. Cerebellar hemorrhage and infarction. Stroke. 1982 Jan-Feb;13(1):106-9. doi: 10.1161/01.str.13.1.106. No abstract available. PMID 7039001
- [Background] Lui TN, Fairholm DJ, Shu TF, Chang CN, Lee ST, Chen HR. Surgical treatment of spontaneous cerebellar hemorrhage. Surg Neurol. 1985 Jun;23(6):555-8. doi: 10.1016/0090-3019(85)90002-3. PMID 3992454
- [Background] Kirollos RW, Tyagi AK, Ross SA, van Hille PT, Marks PV. Management of spontaneous cerebellar hematomas: a prospective treatment protocol. Neurosurgery. 2001 Dec;49(6):1378-86; discussion 1386-7. doi: 10.1097/00006123-200112000-00015. PMID 11846937
- [Background] Datar S, Rabinstein AA. Cerebellar hemorrhage. Neurol Clin. 2014 Nov;32(4):993-1007. doi: 10.1016/j.ncl.2014.07.006. Epub 2014 Sep 11. PMID 25439293
- [Background] Chang CY, Lin CY, Chen LC, Sun CH, Li TY, Tsai TH, Chang ST, Wu YT. The Predictor of Mortality within Six-Months in Patients with Spontaneous Cerebellar Hemorrhage: A Retrospective Study. PLoS One. 2015 Jul 17;10(7):e0132975. doi: 10.1371/journal.pone.0132975. eCollection 2015. PMID 26186721
- [Background] Da Pian R, Bazzan A, Pasqualin A. Surgical versus medical treatment of spontaneous posterior fossa haematomas: a cooperative study on 205 cases. Neurol Res. 1984 Sep;6(3):145-51. doi: 10.1080/01616412.1984.11739680. PMID 6151139
- [Background] van Loon J, Van Calenbergh F, Goffin J, Plets C. Controversies in the management of spontaneous cerebellar haemorrhage. A consecutive series of 49 cases and review of the literature. Acta Neurochir (Wien). 1993;122(3-4):187-93. doi: 10.1007/BF01405527. PMID 8372706
- [Background] Firsching R, Huber M, Frowein RA. Cerebellar haemorrhage: management and prognosis. Neurosurg Rev. 1991;14(3):191-4. doi: 10.1007/BF00310656. PMID 1944934
- [Background] St Louis EK, Wijdicks EF, Li H, Atkinson JD. Predictors of poor outcome in patients with a spontaneous cerebellar hematoma. Can J Neurol Sci. 2000 Feb;27(1):32-6. doi: 10.1017/s0317167100051945. PMID 10676585
- [Background] Lee JH, Kim DW, Kang SD. Stereotactic burr hole aspiration surgery for spontaneous hypertensive cerebellar hemorrhage. J Cerebrovasc Endovasc Neurosurg. 2012 Sep;14(3):170-4. doi: 10.7461/jcen.2012.14.3.170. Epub 2012 Sep 28. PMID 23210043
- [Background] Li L, Li Z, Li Y, Su R, Wang B, Gao L, Yang Y, Xu F, Zhang X, Tian Q, Zhang X, Guo Q, Chang T, Luo T, Qu Y. Surgical Evacuation of Spontaneous Cerebellar Hemorrhage: Comparison of Safety and Efficacy of Suboccipital Craniotomy, Stereotactic Aspiration, and Thrombolysis and Endoscopic Surgery. World Neurosurg. 2018 Sep;117:e90-e98. doi: 10.1016/j.wneu.2018.05.170. Epub 2018 Jun 1. PMID 29864571
- [Background] Meschia JF, Bushnell C, Boden-Albala B, Braun LT, Bravata DM, Chaturvedi S, Creager MA, Eckel RH, Elkind MS, Fornage M, Goldstein LB, Greenberg SM, Horvath SE, Iadecola C, Jauch EC, Moore WS, Wilson JA; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Functional Genomics and Translational Biology; Council on Hypertension. Guidelines for the primary prevention of stroke: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Dec;45(12):3754-832. doi: 10.1161/STR.0000000000000046. Epub 2014 Oct 28. PMID 25355838
- [Background] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Background] Steiner T, Al-Shahi Salman R, Beer R, Christensen H, Cordonnier C, Csiba L, Forsting M, Harnof S, Klijn CJ, Krieger D, Mendelow AD, Molina C, Montaner J, Overgaard K, Petersson J, Roine RO, Schmutzhard E, Schwerdtfeger K, Stapf C, Tatlisumak T, Thomas BM, Toni D, Unterberg A, Wagner M; European Stroke Organisation. European Stroke Organisation (ESO) guidelines for the management of spontaneous intracerebral hemorrhage. Int J Stroke. 2014 Oct;9(7):840-55. doi: 10.1111/ijs.12309. Epub 2014 Aug 24. PMID 25156220
- [Background] Mohadjer M, Eggert R, May J, Mayfrank L. CT-guided stereotactic fibrinolysis of spontaneous and hypertensive cerebellar hemorrhage: long-term results. J Neurosurg. 1990 Aug;73(2):217-22. doi: 10.3171/jns.1990.73.2.0217. PMID 2195140
- [Background] Kellner CP, Moore F, Arginteanu MS, Steinberger AA, Yao K, Scaggiante J, Mocco J, Gologorsky Y. Minimally Invasive Evacuation of Spontaneous Cerebellar Intracerebral Hemorrhage. World Neurosurg. 2019 Feb;122:e1-e9. doi: 10.1016/j.wneu.2018.07.145. Epub 2018 Oct 3. PMID 30292039
- [Background] Khattar NK, Fortuny EM, Wessell AP, John KD, Bak E, Adams SW, Meyer KS, Schirmer CM, Simard JM, Neimat JS, Ding D, James RF. Minimally Invasive Surgery for Spontaneous Cerebellar Hemorrhage: A Multicenter Study. World Neurosurg. 2019 Sep;129:e35-e39. doi: 10.1016/j.wneu.2019.04.164. Epub 2019 Apr 28. PMID 31042595
- [Background] Hackenberg KA, Unterberg AW, Jung CS, Bosel J, Schonenberger S, Zweckberger K. Does suboccipital decompression and evacuation of intraparenchymal hematoma improve neurological outcome in patients with spontaneous cerebellar hemorrhage? Clin Neurol Neurosurg. 2017 Apr;155:22-29. doi: 10.1016/j.clineuro.2017.01.019. Epub 2017 Feb 3. PMID 28226284
- [Background] Lee TH, Huang YH, Su TM, Chen CF, Lu CH, Lee HL, Tsai HP, Sung WW, Kwan AL. Predictive Factors of 2-Year Postoperative Outcomes in Patients with Spontaneous Cerebellar Hemorrhage. J Clin Med. 2019 Jun 8;8(6):818. doi: 10.3390/jcm8060818. PMID 31181777
- [Background] Al Safatli D, Guenther A, McLean AL, Waschke A, Kalff R, Ewald C. Prediction of 30-day mortality in spontaneous cerebellar hemorrhage. Surg Neurol Int. 2017 Nov 20;8:282. doi: 10.4103/sni.sni_479_16. eCollection 2017. PMID 29279799
- [Background] Liu H, Wu X, Tan Z, Guo H, Bai H, Wang B, Cui W, Zheng L, Sun F, Zhang X, Fan R, Wang P, Jing W, Gao J, Guo W, Qu Y. Long-Term Effect of Endoscopic Evacuation for Large Basal Ganglia Hemorrhage With GCS Scores <== 8. Front Neurol. 2020 Aug 14;11:848. doi: 10.3389/fneur.2020.00848. eCollection 2020. PMID 32922354
- [Background] Guo W, Liu H, Tan Z, Zhang X, Gao J, Zhang L, Guo H, Bai H, Cui W, Liu X, Wu X, Luo J, Qu Y. Comparison of endoscopic evacuation, stereotactic aspiration, and craniotomy for treatment of basal ganglia hemorrhage. J Neurointerv Surg. 2020 Jan;12(1):55-61. doi: 10.1136/neurintsurg-2019-014962. Epub 2019 Jul 12. PMID 31300535